CLINICAL TRIAL: NCT05739136
Title: MYFEMBREE®: A Retrospective Cohort Study Using an Administrative Healthcare Database to Assess Pregnancy Outcomes in Women Treated With Relugolix Combination Therapy
Status: Active, not recruiting | Type: Observational
Sponsor: Sumitomo Pharma Switzerland GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: MVT-601A-003
Record Dates: First submitted 2023-02-13; First posted 2023-02-22 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Pregnancy Related; Pregnancy Complications; Pregnancy, High Risk
Keywords: Relugolix; Uterine Fibroids; Endometriosis; Pregnancy
MeSH Terms: conditions — Pregnancy Complications; Leiomyoma; Endometriosis | interventions — relugolix; Estradiol; Norethindrone Acetate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Exposed Cohort: Pregnant women with conditions for which relugolix combination therapy is prescribed, who are exposed to relugolix combination therapy at any time during pregnancy
  Interventions: Drug: Relugolix + Estradiol + Norethindrone Acetate
- Unexposed Cohort: Pregnant women with conditions for which relugolix combination therapy could be prescribed, who are not exposed to relugolix combination therapy at any time during pregnancy

INTERVENTIONS:
Drug: Relugolix + Estradiol + Norethindrone Acetate — Relugolix combination therapy (relugolix 40 mg; estradiol 1 mg; norethindrone 0.5 mg)
  Other Names: MVT-601; MVT-601A; MYFEMBREE
  Groups: Exposed Cohort

SUMMARY:
This is a retrospective cohort study that will be conducted using secondary de-identified electronic healthcare data (EHD) that originally were collected for the purposes of health insurance billing and/or routine patient care from healthcare providers (HCPs). The study is designed to evaluate the association between relugolix combination therapy (relugolix 40 mg, estradiol 1 mg, and norethindrone acetate 0.5 mg) exposure during pregnancy and subsequent fetal and infant outcomes.

DETAILED DESCRIPTION:
The study will identify pregnant women exposed to relugolix combination therapy during pregnancy from a United States (US) administrative claims database. The primary outcome measure is major congenital malformations (MCMs) among linked live births. Secondary outcome measures include spontaneous abortion (SAB), stillbirth, small size for gestational age (SGA), and preterm birth. Infants of pregnancies with linked live birth outcomes will be followed up to 12 months of age for identification of MCMs. Anticipated enrollment is 530 live births.

ELIGIBILITY:
Inclusion Criteria:

* Woman ≥ 18 and ≤ 50 years of age at time of conception
* Diagnosis of a condition for which relugolix combination therapy is prescribed (diagnosis captured at any time prior to the estimated date of conception)

Cohort 1

* Exposure to relugolix combination therapy at any time during pregnancy

Cohort 2

* No exposure to relugolix combination therapy at any time after the estimated date of conception (during pregnancy)

Exclusion Criteria:

* Exposure to known teratogens during pregnancy
* < 6 months of continuous healthcare coverage immediately prior to date of conception

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: The study population will include 2 cohorts: The exposed cohort will include pregnant women with conditions for which relugolix combination therapy is prescribed and who are exposed to relugolix combination therapy at any time during pregnancy. The unexposed cohort will include pregnant women with conditions for which relugolix combination therapy could be prescribed and who are not exposed to relugolix combination therapy at any time during pregnancy.
Sampling Method: Non-Probability Sample
Enrollment: 530 (Estimated)
Dates: Start 2025-04-30 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Major Congenital Malformation (MCM) | Up to 5 years
  Comparison of rate of MCM between cohorts

SECONDARY OUTCOMES:
Spontaneous abortion (SAB) | Up to 5 years
  Comparison of rate of SABs between cohorts
Stillbirth | Up to 5 years
  Comparison of rate of stillbirths between cohorts
Preterm birth | Up to 5 years
  Comparison of rate of preterm births between cohorts
Small for gestational age (SGA) | Up to 5 years
  Comparison of rate of SGA between cohorts

CONTACTS AND LOCATIONS:
Locations (1):
- SMPA, Marlborough, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No